CLINICAL TRIAL: NCT03536663
Title: An Open-Label Clinical Study to Assess the Performance of the Dialyzer With Endexo™ in End-Stage Renal Disease Subjects
Brief Title: Clinical Study to Assess the Performance of the Dialyzer With Endexo™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care North America (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Endexo-001
Record Dates: First submitted 2018-04-06; First posted 2018-05-25 (Actual); Results first posted 2020-11-12 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: 12 HD treatments (4 weeks) with Optiflux dialyzer followed by 38 HD treatments (13 weeks) with Endexo dialyzer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Optiflux/Endexo (Other): Optiflux (Active Comparator); Hemodialysis treatments on the Optiflux dialyzer (Optiflux Period) for 4 weeks - Visit 1 to 12 Endexo (Experimental); Subjects continue on Dialyzer with Endexo (Endexo Period) for 13 weeks - Visit 13 to visit 50
  Interventions: Device: Optiflux and Dialyzer with Endexo

INTERVENTIONS:
Device: Optiflux and Dialyzer with Endexo — Hemodialysis (HD) on Optiflux dialyzer from Visit 1 to 12 and followed by HD on the dialyzer with Endexo at visit 13 and continues until visit 50. Dialysis is performed 3 times per week which means the total of the intervention will be 17 weeks.

SUMMARY:
Endexo™ is an additive that is blended into the fiber solution during manufacturing of the hemodialyzer hollow fibers. The intended purpose of the additive is to increase blood compatibility in the finished dialyzer, which is referred to as the "dialyzer with Endexo."

DETAILED DESCRIPTION:
This is a prospective, sequential, multi-center, open-label study with subjects on thrice-weekly (in-center) hemodialysis (HD). After a Screening Period, there will be 12 hemodialysis treatments on the Optiflux dialyzer (Optiflux Period), followed by 38 HD treatments on the dialyzer with Endexo (Endexo Period), and then a Follow-up Visit. The study population will consist of End-Stage Renal Disease ESRD subjects who are a minimum of 22 years of age. The primary objective of the study is to collect data on the performance of the dialyzer with Endexo when used to perform hemodialysis (HD) in End-Stage Renal Disease (ESRD) subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Must be an adult, older than 22 years of age.
2. Has been prescribed in-center thrice-weekly HD continuously for at least 180 days prior to the date of signed informed consent
3. Has been prescribed the Optiflux F160NR dialyzer continuously for at least 30 days prior to the date of signed informed consent
4. Has a prescribed HD treatment time ≥180 minutes (3 hours) and ≤270 minutes (4.5 hours)
5. Has been on heparin anticoagulation for dialysis and has had no change in heparin prescription within 14 days prior to the date of signed informed consent
6. Has a most recent single pool Kt/V (spKt/V) ≥1.2 within 45 days prior to the date of a signed informed consent
7. Has a most recent hemoglobin ≥9 g/dL within 45 days prior to the date of a signed informed consent
8. Has a most recent platelet count ≥100,000/mm3 within 45 days prior to the date of a signed informed consent
9. A female of childbearing potential must have a negative serum pregnancy test at the time of screening and agree to use an acceptable method of contraception during the study

Exclusion Criteria:

1. Use of citric acid concentrate (such as Citrasate®) at the time of signed informed consent
2. Known allergic reactions to Endexo
3. Hospitalization within 30 days prior to the date of signed informed consent
4. Presence of active malignancy, congestive heart failure New York Heart Association (NYHA) Class III or IV, or liver cirrhosis
5. Are receiving or have received chemotherapy / radiation therapy / plasmapheresis therapy within 90 days prior to the date of signed informed consent
6. Are receiving antibiotics or have used antibiotics within 14 days prior to the date of signed informed consent
7. Are currently enrolled in or have completed any other investigational product study within 30 days prior to the date of signed informed consent
8. Has a life expectancy of less than 1 year

Ages: 22 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shakil Aslam, MD, Study Director — Fresenius Medical Care RTG, LLC; Dylan Steer, MD, Principal Investigator — California Institute of Renal Research; Lisa Weber, MD, Principal Investigator — Research Management Inc/ Kansas Nephrology Research Institute, LLC-J/V; Jill Meyer, MD, Principal Investigator — Balboa Nephrology Med Group
Locations (3):
- United States (3):
  - Balboa Nephrology Med Group, Chula Vista, California
  - California Institute of Renal Research, San Diego, California
  - Research Management Inc/ Kansas Nephrology Research Institute, LLC-J/V, Wichita, Kansas

REFERENCES:
- [Derived] Meyer JM, Steer D, Weber LA, Zeitone AA, Thakuria M, Ho CH, Aslam S, Mullon C, Kossmann RJ. Safety of a Novel Dialyzer Containing a Fluorinated Polyurethane Surface-Modifying Macromolecule in Patients with End-Stage Kidney Disease. Blood Purif. 2021;50(6):959-967. doi: 10.1159/000514937. Epub 2021 Mar 31. PMID 33789265

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hemodialysis patients were recruited at three clinical sites in the USA. 23 subjects were enrolled to this study. The first subject first visit was on August 29, 2018 and the last subject last visit was on April 17, 2019.
Groups:
- Optiflux/Endexo: Hemodialysis treatments on the dialyzer with Endexo starts at visit 13 and continues until visit 50. Dialysis is performed 3 times per week which means the total of the intervention is approximately 12 weeks.
  Dialyzer with Endexo: Hemodialysis treatments on the dialyzer with Endexo starts at visit 13 and continues until visit 50. Dialysis is performed 3 times per week which means the total of the intervention is approximately 12 weeks.
Period: Optiflux
Arm/Group | Optiflux/Endexo
Started | 23
Completed | 19
Not Completed | 4
Period: Endexo
Arm/Group | Optiflux/Endexo
Started | 18 (One subject completed the Optiflux period but missed Visit 13 and was withdrawn per protocol.)
Completed | 17
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Subjects who sign the ICF, are eligible, are enrolled in the study, and have at least one HD treatment with the dialyzer with Endexo.
Groups:
- Endexo: Hemodialysis treatments on the dialyzer with Endexo starts at visit 13 and continues until visit 50. Dialysis is performed 3 times per week which means the total of the intervention is approximately 13 weeks.
  Dialyzer with Endexo: Hemodialysis treatments on the dialyzer with Endexo starts at visit 13 and continues until visit 50. Dialysis is performed 3 times per week which means the total of the intervention is approximately 13 weeks.
Arm/Group | Endexo
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.28 (14.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 12
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Performance of the Dialyzer With Endexo by Measuring Its in Vivo Ultrafiltration Coefficient
Description: Ultrafiltration coefficient (Kuf) is the ratio of ultrafiltration rate in ml/hr to the Transmembrane pressure in mmHg. Both the Ultrafiltration rate and the transmembrane pressure readings are collected from the machine.
Time Frame: 15 minutes after the recorded start of hemodialysis with Endexo upon its first use in the study
Population: Subjects who are in the safety population, and have a minimum of 36 HD treatments with the dialyzer with Endexo.
Measure: Mean (Standard Deviation); unit: mL/hr/mmHg
Groups:
- Endexo: Hemodialysis treatments on the dialyzer with Endexo starts at visit 13 and continues until visit 50. Dialysis is performed 3 times per week which means the total of the intervention will be 13 weeks.
  Dialyzer with Endexo: Hemodialysis treatments on the dialyzer with Endexo starts at visit 13 and continues until visit 50. Dialysis is performed 3 times per week which means the total of the intervention will be 13 weeks.
Arm/Group | Endexo
Number analyzed (Participants) | 17
mL/hr/mmHg | 16.36 (9.92)

2. Secondary Outcome: The Number of Any Adverse Events
Description: All adverse events were captured from subject enrollment to the completion of Optiflux period, and to the end of study or withdraws from the study.
Time Frame: Optiflux: from enrollment, weeks 1 to 4 (visits 1 to 12); Endexo: from weeks 5 to 17, and follow-up, a total of 17 weeks intervention.
Population: Subjects who sign the ICF, are eligible, are enrolled in the study for Optiflux, and have at least one HD treatment with Endexo dialyzer for Endexo.
Measure: Number; unit: events
Groups:
- Optiflux: Optiflux dialyzer: Hemodialysis treatments on the optiflux dialyzer starts at visit 1 and continues until visit 12.
- Endexo: Dialyzer with Endexo: Hemodialysis treatments on the dialyzer with Endexo starts at visit 13 and continues until visit 50.
Arm/Group | Optiflux | Endexo
Number analyzed (Participants) | 23 | 18
events | 7 | 32

3. Secondary Outcome: The Number of Any Device-related Adverse Events
Description: Any device-related adverse events were captured from subject enrollment to the completion of Optiflux period, and to the end of study or withdraws from the study.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: participants, events
Groups:
- Optiflux: Optiflux d: Hemodialysis treatments on the dialyzer with Endexo starts at visit 1 and continues until visit 12.
Arm/Group | Optiflux | Endexo
Number analyzed (Participants) | 23 | 18
participants, events | 0 | 0

4. Secondary Outcome: Removal of Urea
Description: 1. URR = (pre-HD urea - post-HD urea)/pre-HD urea * 100
  2. Data across visits were averaged for each subject, and then a group mean and sd were calculated.
Time Frame: At visits 1/week 1, 10/week 4, 13/week 5, 22/week 8, 34/week 12, and 46/week 16
Population: Subjects who are in the safety population, and have a minimum of 36 HD treatments with the dialyzer with Endexo.
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Optiflux: Optiflux dialyzer: Hemodialysis treatments on the dialyzer with Endexo starts at visit 1 and continues until visit 12.
Arm/Group | Optiflux | Endexo
Number analyzed (Participants) | 17 | 17
percentage | 80.81 (4.33) | 81.87 (5.91)

5. Secondary Outcome: Removal of Albumin
Description: %change = (post-HD - pre-HD)/pre-HD * 100
Time Frame: Pre- and Post- HD at Visits 1/week 1, 13/week 5
Population: Subjects who are in the safety population, and have a minimum of 36 HD treatments with the dialyzer with Endexo.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Optiflux | Endexo
Number analyzed (Participants) | 17 | 17
percent change | 7.89 (8.63) | 7.99 (7.25)

6. Secondary Outcome: Removal of Beta-2-microglobulin
Description: % reduction = (post-HD - pre-HD)/pre-HD * 100 with post-HD B2M adjusted to pre- and post HD weights
Time Frame: Pre- and Post- HD at Visits 1/week 1, 13/week 5
Population: Subjects who are in the safety population, and have a minimum of 36 HD treatments with the dialyzer with Endexo.
  One subject in this pop did not have lab results for pre- and post beta-2-microglobulin in Endexo period. Therefore n=16 instead of 17.
Measure: Mean (Standard Deviation); unit: percent reduction, corrected
Arm/Group | Optiflux | Endexo
Number analyzed (Participants) | 17 | 16
percent reduction, corrected | 46.86 (7.16) | 67.73 (16.32)

7. Other Pre Specified Outcome: Dialyzer Hemocompatibility
Description: The dialyzer hemo-compatibility is measured by measuring the activation of the complement system (C3a, C5a, SC5b-9)
Time Frame: Assessed at the first time the dialyzers are used in the study , collected pre hemodialysis and 30 minutes after the recorded start of hemodialysis
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Clotting of the Dialyzer
Description: Thrombus scoring will be assessed according to a clotting scale (The graded scoring method)
Time Frame: visual evaluation of the dialyzer arterial cap will be performed at the end of every hemodialysis treatment to determine the Grade:1,2,3 or 4. (1:no clotting to 4: total clotting), throughout a total of 17 weeks intervention.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: a max of 22 weeks for a subject to complete the study
Groups:
- Optiflux: Hemodialysis treatments on Optiflux dialyzer starts at visit 1 and continues for 4 weeks to visit 12. Dialysis is performed 3 times per week which means the total of the intervention will be 13 weeks.
- Endexo: Hemodialysis treatments on the dialyzer with Endexo starts at visit 13 and continues until visit 50. Dialysis is performed 3 times per week which means the total of the intervention will be 13 weeks.
Arm/Group | Optiflux | Endexo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/23 | 3/18
Other Adverse Events (participants affected / at risk) | 4/23 | 11/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optiflux (N=23) | Endexo (N=18)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | NA | 1 (1) — GASTROINTESTINAL BLEEDING
Localised infection (Infections and infestations) | NA | 1 (1) — RIGHT FOOT INFECTION
Hypertensive emergency (Vascular disorders) | NA | 1 (1) — HYPERTENSIVE EMERGENCY
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optiflux (N=23) | Endexo (N=18)
Orbital oedema (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bowel movement irregularity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 2 (2)
Tissue infiltration (General disorders) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT03536663/SAP_000.pdf
  • Study Protocol (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT03536663/Prot_001.pdf